CLINICAL TRIAL: NCT04127643
Title: Prospective Clinical Registry of Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) (S-ICD Korea Registry)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2019-0022
Record Dates: First submitted 2019-10-08; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure; Sudden Cardiac Death; Ventricular Tachycardia
Keywords: S-ICD; safety; feasibility
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- S-ICD patients: patients who have received the EMBLEM S-ICD system

SUMMARY:
S-ICD avoids the use intravascular leads and their associated risks, has been increasingly used for primary and secondary prevention of sudden death. The long-term safety and feasible of S-ICD system in Asian population with a smaller body size remain unclear. The investigators propose to perform a prospective study in Korean population to investigate the safety and feasibility of S-ICD for primary or secondary prevention of sudden cardiac death.

DETAILED DESCRIPTION:
The investigators propose to prospectively recruit 300 patients who are qualified to receive the EMBLEM S-ICD system by following the proposed BSC Patient Screening Steps in 10 sites in Korea. All patients will be follow-up as standard of care to collect acute procedural and device related complications as well as long-term, device related, clinical and patient reported outcomes. Follow up data will be systematically collected over 24 months post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Patients with conventional indications for ICD and;
3. Ability to provide informed consent and to complete the study and required follow-up

Exclusion Criteria:

1. planned cardiac surgery within 3 months of enrollment;
2. pregnancy;
3. life expectancy <3 months;
4. indication for CRT-D or permanent ventricular pacing for new implant;
5. incessant ventricular tachycardia and/or spontaneous, frequently recurring ventricular tachycardia that is reliably terminated with anti-tachycardia pacing; and
6. patients with unipolar pacemakers or implanted devices that revert to unipolar pacing

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have received the EMBLEM S-ICD system
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Perioperative S-ICD Complication Free Rate up to 7 days post implant | 7 days
Perioperative S-ICD Complication Free Rate up to 30 days post implant | 30 days
1 year S-ICD Complication Free Rate | 1 year
2 year S-ICD Complication Free Rate | 2 year
Percentage of inappropriate shocks for AF/SVT | 7 days
Percentage of inappropriate shocks for AF/SVT | 30 days
Percentage of inappropriate shocks for AF/SVT | 1 year
Percentage of inappropriate shocks for AF/SVT | 2 year

SECONDARY OUTCOMES:
Device related discomfort | 7 days
  Device related discomfort means pain, the limitation of movement of body or any discomfort reported by the patients.
Device related discomfort | 30 days
  Device related discomfort means pain, the limitation of movement of body or any discomfort reported by the patients.
Device related discomfort | 1 year
  Device related discomfort means pain, the limitation of movement of body or any discomfort reported by the patients.
Device related discomfort | 2 year
  Device related discomfort means pain, the limitation of movement of body or any discomfort reported by the patients.
Efficacy of S-ICD therapy for spontaneous VT/VF | 7 days
  Efficacy of S-ICD therapy for spontaneous VT/VF means the successful termination of spontaneous VT/VF by the shock delivered by S-ICD therapy.
Efficacy of S-ICD therapy for spontaneous VT/VF | 30 days
  Efficacy of S-ICD therapy for spontaneous VT/VF means the successful termination of spontaneous VT/VF by the shock delivered by S-ICD therapy.
Efficacy of S-ICD therapy for spontaneous VT/VF | 1 year
  Efficacy of S-ICD therapy for spontaneous VT/VF means the successful termination of spontaneous VT/VF by the shock delivered by S-ICD therapy.
Efficacy of S-ICD therapy for spontaneous VT/VF | 2 year
  Efficacy of S-ICD therapy for spontaneous VT/VF means the successful termination of spontaneous VT/VF by the shock delivered by S-ICD therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No